CLINICAL TRIAL: NCT03469167
Title: Clinical Study to Evaluate Efficacy and Safety of "CEGP003(Wound Dressing Solution Containing EGF)" for Achieving Hemostasis and Protecting Ulcer in Patients With Acute Peptic Ulcer Bleeding: A Prospective, Randomized Trial
Brief Title: Study to Evaluate Efficacy and Safety of Wound Dressing Solution Containing EGF in Patients With Peptic Ulcers Bleeding
Acronym: CEGP003
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CGBio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CGB-01
Record Dates: First submitted 2018-03-05; First posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Peptic Ulcer Bleeding
Keywords: Bleeding
MeSH Terms: conditions — Peptic Ulcer Hemorrhage; Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CEGP003 (Experimental)
  Interventions: Device: CEGP003
- Injection Tx (Active Comparator)
  Interventions: Device: Injection Tx

INTERVENTIONS:
Device: CEGP003 — Application of CEGP003 to peptic ulcer bleeding
  Other Names: EGF
  Arms: CEGP003
Device: Injection Tx — Injection of epinephrine to peptic ulcer bleeding
  Other Names: epinephrine injection
  Arms: Injection Tx

SUMMARY:
This is a prospective, single-blinded, randomized study to evaluate the efficacy and safety of CEGP003 in patients with acute peptic ulcers bleeding, compared to endoscopic epinephrine injection therapy.

DETAILED DESCRIPTION:
CEGP003 is wound dressing solution containing Hydroxyethyl-cellulose and EGF. Epidermal growth factor (EGF) stimulates cell growth and differentiation by binding to its receptor, which can enhance wound healing and regeneration of new tissue, finally may provide a new option in treating a peptic ulcers bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Peptic ulcer with high-risk stigmata of recent hemorrhage (Forrest class IA, IB, IIA and IIB)

Exclusion Criteria:

* Subjects who have a history of malignant tumor in upper gastro-intestinal site
* Subjects with platelet and coagulation dysfunction (PLT < 50E9/L, INR > 2)
* Subjects that have taken anticoagulant drugs or non-steroidal anti-inflammatory drugs within 72 hours after the treatment
* Subjects with one or more bleeding sources
* Subjects who are pregnant or breast-feeding
* Subject who are allergic or have a hypersensitive reaction to Hydroxyethyl-cellulose or EGF
* Subjects who have undergone endoscopically therapies within the last 7 days
* Subjects who are considered not suitable for the study by significant disease
* Subjects who are not able to comply with the study requirements
* Subjects who are currently enrolled in another clinical study which can impact the study within 30 days of screening
* Subjects who are considered not suitable for the study by the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-10-15 (Actual); Primary Completion 2015-11-10 (Actual); Study Completion 2017-01-02 (Actual)

PRIMARY OUTCOMES:
Initial hemostasis rate | Within 10 minutes after first endoscopy session
  Endoscopically verified cessation of bleeding for at least 10 minutes after treatment.

SECONDARY OUTCOMES:
Recurrent bleeding rate | Within 72 hours
  If any of the following conditions are met, an endoscopy will verify for rebleeding.
  * Associated with overt signs of GI bleed (melena, and/or hematemesis)
  * Instability of Vital signs (<80/60 mmHg of blood pressure, and/or >120 beats/min of pulse)
  * Decrease in hemoglobin of at least 2 g/dl after Initial hemostasis
  * bleeding can be confirmed directly (direct visualization)
Time required for treatment | 0 day
  The time from when the endoscope is inserted to when the endoscope treatment is completed.
Wound healing effect of peptic ulcer | After 3 days (72 hours)
  Evaluation of Stage Classification of Gastric Ulcer by Sakita-Miwa.
Usability for the delivery system | 0 day
  Evaluation of success for the delivery system

CONTACTS AND LOCATIONS:
Overall Officials: Don Haeng Lee, MD. PhD., Principal Investigator — Inha University Hospital; Su Jin Hong, MD. PhD., Principal Investigator — Soon Chun Hyang University

IPD SHARING:
Plan to Share IPD: No